CLINICAL TRIAL: NCT01395030
Title: Genomic and Imaging Study for Patients Undergoing Surgery for Liver Cancer
Brief Title: PET/CT in Diagnosing Patients With Liver Cancer Undergoing Surgical Resection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Queen's Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Sandi Kwee, Principal Investigator, Queen's Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RA-2011-025; NCI-2012-02095 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CHS-19373 (Other: University of Hawaii); RA-2011-025 (Other: Queen's Medical Center); R01CA161209 (NIH)
Record Dates: First submitted 2011-07-12; First posted 2011-07-15 (Estimated); Results first posted 2018-09-26 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-08

CONDITIONS: Adult Hepatocellular Carcinoma; Localized Resectable Adult Liver Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Tomography, X-Ray Computed; Tomography; fluoromethylcholine; fluorocholine; Positron-Emission Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 18F-fluoromethylcholine PET/CT (Experimental): Patients undergo 18F-fluoromethylcholine positron emission tomography (PET)/ computed tomography (CT) scan within 14 days of surgical resection of liver tumor.
  Interventions: Diagnostic Test: Computed Tomography; Drug: 18F-fluoromethylcholine; Diagnostic Test: Positron Emission Tomography

INTERVENTIONS:
Diagnostic Test: Computed Tomography — Undergo FCH PET/CT
  Other Names: Computerized Axial Tomography; computerized tomography; CT; CT scan; tomography
Drug: 18F-fluoromethylcholine — Undergo FCH PET/CT
  Other Names: fluorine-18 fluoromethylcholine; 18F-fluorocholine; 18F-choline; FCH
Diagnostic Test: Positron Emission Tomography — Undergo FCH PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This clinical trial studies positron emission tomography (PET)/computed tomography (CT) in diagnosing patients with liver cancer undergoing surgical resection. Diagnostic procedures, such as fluorine-18 fluoromethylcholine PET/CT, may help find and diagnose liver cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the most optimal fluorine-18 (18F) fluoromethylcholine (FCH) PET/CT parameters for detecting primary hepatocellular carcinoma (HCC) by conducting a clinical radiologic-pathologic correlation study to estimate and compare the receiver operating characteristics of kinetic and static PET measures of tumor FCH metabolism in patients that test positive during screening or conventional imaging.

II. Identify cancer signaling pathways associated with choline metabolism in HCC by profiling the global gene expression patterns in fresh-frozen liver tissue samples that are correlated with the features derived from FCH PET/CT images.

III. Characterize the association between features derived from FCH PET/CT images of the liver and clinical liver disease severity and comparatively evaluate the ability of corresponding gene expression signatures to predictively model HCC disease outcome.

OUTLINE:

Patients undergo 18F-fluoromethylcholine PET/CT within 14 days of surgical resection.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Liver tumor diagnosed histologically as HCC or suspected of being HCC in association with serum alpha-fetoprotein level > 200 or tumor mass with characteristics of malignancy on diagnostic imaging
* Under the care of a surgical attending
* Deemed a surgical candidate and has agreed to surgery to remove a portion of the liver containing tumor
* Child-Pugh A/B

Exclusion Criteria:

* Weight > 350 lbs
* Pregnant or lactating female, a serum pregnancy test will be performed within 2 weeks or less before the date of the FCH PET/CT scan in all women capable of becoming pregnant
* Serious underlying medical condition that would impair patient's ability to tolerate the imaging procedure
* Concurrent treatment with chemotherapy, molecule-selective, biological, or radiotherapeutic agent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2011-08-15 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2018-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandi Kwee, MD, Principal Investigator — Queen's Medical Center
Locations (1):
- University of Hawaii Cancer Center, Honolulu, Hawaii, United States

REFERENCES:
- [Result] Kwee SA, Wong L, Chan OTM, Kalathil S, Tsai N. PET/CT with 18F Fluorocholine as an Imaging Biomarker for Chronic Liver Disease: A Preliminary Radiopathologic Correspondence Study in Patients with Liver Cancer. Radiology. 2018 Apr;287(1):294-302. doi: 10.1148/radiol.2018171333. Epub 2018 Jan 9. PMID 29315063

RESULTS

PARTICIPANT FLOW:
Groups:
- 18F-fluoromethylcholine PET/CT: Patients undergo fluorine-18 (18F-) fluoromethylcholine (FCH) positron emission tomography (PET)/ computed tomography (CT) scan within 14 days of surgical resection.
  Computed Tomography: Undergo FCH PET/CT
  18F-fluoromethylcholine: Undergo FCH PET/CT
  Laboratory Biomarker Analysis: Correlative studies
  Positron Emission Tomography: Undergo FCH PET/CT
Period: Overall Study
Arm/Group | 18F-fluoromethylcholine PET/CT
Started | 64
Complete FCH PET/CT | 57
Adequate Tissue for Analysis | 50
Completed | 57
Not Completed | 7
Not completed — Did not complete FCH PET/CT | 7

BASELINE CHARACTERISTICS:
Population: Study subjects who completed FCH PET/CT
Groups:
- 18F-fluoromethylcholine PET/CT: Patients undergo 18F-fluoromethylcholine PET/CT scan within 14 days of surgical resection.
  Computed Tomography: Undergo FCH PET/CT
  18F-fluoromethylcholine: Undergo FCH PET/CT
  Laboratory Biomarker Analysis: Correlative studies
  Positron Emission Tomography: Undergo FCH PET/CT
Arm/Group | 18F-fluoromethylcholine PET/CT
Number analyzed (Participants) | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 37
  >=65 years | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 56
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 29
  Native Hawaiian or Other Pacific Islander | 13
  Black or African American | 2
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 57
Tumor Diagnosis [Count of Participants; unit: Participants]
  Hepatocellular carcinoma | 48
  Cholangiocarcinoma | 8
  Sarcoma | 1

OUTCOME MEASURES:

1. Primary Outcome: Fluorine-18 (18F) Fluoromethylcholine (FCH) PET/CT Parameters for Assessing Hepatocellular Carcinoma (HCC): Area Under the Receiver Operating Characteristic Curve.
Description: Area under the receiver operating characteristic curve for detecting resectable hepatocellular carcinoma with prognostically favorable molecular features (Hoshida molecular sub-class S3) based on FCH PET/CT measurement of tumor maximum standardized uptake value (SUVmax).
Time Frame: Up to study completion at an average of 2.5 years
Population: Patients from whom surgical tumor resection (ie. partial hepatectomy) provided adequate tumor and liver samples for tissue analysis.
Measure: Number; unit: unitless
Arm/Group | 18F-fluoromethylcholine PET/CT
Number analyzed (Participants) | 50
unitless
  All primary liver cancers (n=50) | 0.87
  HCC only (n=41): number analyzed (Participants) | 41
  HCC only (n=41) | 0.80

2. Primary Outcome: Fluorine-18 (18F) Fluoromethylcholine (FCH) PET/CT Parameters for Assessing Hepatocellular Carcinoma (HCC): Sensitivity/Specificity
Description: Sensitivity and specificity estimated at a predefined point (ie. Youden's maxima) on the receiver operating characteristic curve for detecting hepatocellular carcinoma with prognostically favorable molecular features (Hoshida molecular sub-class S3) based on FCH PET/CT measurement of tumor maximum standardized uptake value (SUVmax) in patients who underwent subsequent tumor resection.
Time Frame: Up to study completion at an average of 2.5 years
Population: as for outcome 1
Measure: Number; unit: percentage of analyzed participants
Arm/Group | 18F-fluoromethylcholine PET/CT
Number analyzed (Participants) | 50
percentage of analyzed participants
  Sensitivity for HCC sub-class S3 | 100
  Specificity for HCC sub-class S3 | 73

3. Primary Outcome: Statistical Significance of Molecular Pathways Associated With Choline Metabolism as Identified Through Gene Set Enrichment Analysis of Hepatocellular Carcinoma (HCC) Tumor Samples.
Description: Statistically significant enrichment by sets of genes corresponding to previously-defined molecular pathway signatures was assessed by gene set enrichment analysis (a publicly available algorithm) of whole-genome expression array data obtained from tumors previously characterized by FCH PET/CT. Statistical significance was based on a false discovery rate < 0.05. Tumors demonstrating high choline metabolism (defined by a tumor-liver ratio > 1.0 measured on PET) were assessed for enrichment by publicly-available gene sets. This particular analysis involved the entire Molecular Hallmarks gene signature collection (v6.0) as obtained from the Broad Institute Molecular Signature Database (MSigDB).
Time Frame: Up to study completion at an average of 2.5 years
Population: Patients with histopathologically confirmed HCC who completed FCH PET/CT followed by completion of whole-genome expression array analysis of tumor and adjacent liver tissue obtained following partial hepatectomy.
Measure: Number; unit: false discovery rate
Arm/Group | 18F-fluoromethylcholine PET/CT
Number analyzed (Participants) | 41
false discovery rate
  HALLMARK_OXIDATIVE_PHOSPHORYLATION | 0.009
  HALLMARK_ADIPOGENESIS | 0.012
  HALLMARK_PEROXISOME | 0.012
  HALLMARK_XENOBIOTIC_METABOLISM | 0.014
  HALLMARK_FATTY_ACID_METABOLISM | 0.015
  HALLMARK_BILE_ACID_METABOLISM | 0.016
Statistical Analysis 1: Comparison: 18F-fluoromethylcholine PET/CT; Test type: Other; Analysis was performed using Gene Set Enrichment Analysis (GSEA version 19.0.24, Broad Institute, Cambridge, MA) implemented in GenePattern (Broad Institute, Cambridge, MA) by uploading expression array data to this cloud-computing genomics platform. The specific details of this statistical approach can be found in the following publicly available references: Reich M, Liefeld T, Gould J, Lerner J, Tamayo P, Mesirov JP. GenePattern 2.0 Nature Genetics 38 no. 5 (2006): pp500-501 Subramanian A, Tamayo P, Mootha VK, Mukherjee S, Ebert BL, Gillette MA, Paulovich A, Pomeroy SL, Golub TR, Lander ES, Mesirov JP. Gene set enrichment analysis: A knowledge-based approach for interpreting genome-wide expression profiles. PNAS. 2005;102(43);15545-15550

4. Primary Outcome: Clinical Liver Disease Severity Based on Liver Fibrosis (Metavir) Stage
Description: Odds ratios and 95% confidence intervals for histologic liver fibrosis (Metavir) stage >= F1, >= F2, >= F3, and F4 at liver standardized uptake value (SUV) thresholds of 8.3, 8.0, 7.4, and 6.4, respectively. Reference: PMID 29315063.
Time Frame: Up to 1 year
Population: Number of subjects with available peri-tumoral liver histopathology data
Measure: Number (95% Confidence Interval); unit: odds ratio
Arm/Group | 18F-fluoromethylcholine PET/CT
Number analyzed (Participants) | 48
odds ratio
  Fibrosis stage >= F1 | 3.03 [1.59 to 5.88]
  Fibrosis stage >= F2 | 5.29 [1.79 to 7.69]
  Fibrosis stage >= F3 | 5.56 [1.85 to 16.7]
  Fibrosis stage F4 | 6.67 [1.33 to 33.3]

5. Primary Outcome: Number of Participants Comprising Two Distinct PET/CT Imaging Phenotypes (High FCH Uptake vs. Low FCH Uptake) Between the Different Tumor Sub-classes
Description: HCC tumors were sub-classified using gene expression arrays into 3 distinct prognostically-relevant molecular sub-classes (S1,S2, S3, where S3 is associated with the most favorable clinical prognosis) based on Hoshida et. al (PMID 19723656). The number of tumors comprising two distinct PET/CT imaging phenotypes (high FCH uptake vs. low FCH uptake) was compared between the different sub-classes.
Time Frame: Up to study completion at an average of 2.5 years
Population: Patients who underwent FCH PET/CT followed by histopathologic confirmation of the tumor
Measure: Count of Participants; unit: Participants
Arm/Group | 18F-fluoromethylcholine PET/CT
Number analyzed (Participants) | 50
Participants
  HCC sub-class S1: number analyzed (Participants) | 13
  HCC sub-class S1: High FCH uptake | 7
  HCC sub-class S1: Low FCH uptake | 6
  HCC sub-class S2: number analyzed (Participants) | 4
  HCC sub-class S2: High FCH uptake | 0
  HCC sub-class S2: Low FCH uptake | 4
  HCC sub-class S3: number analyzed (Participants) | 24
  HCC sub-class S3: High FCH uptake | 24
  HCC sub-class S3: Low FCH uptake | 0
  Intrahepatic cholangiocarcinoma: number analyzed (Participants) | 8
  Intrahepatic cholangiocarcinoma: High FCH uptake | 0
  Intrahepatic cholangiocarcinoma: Low FCH uptake | 8
  Primary sarcoma: number analyzed (Participants) | 1
  Primary sarcoma: High FCH uptake | 0
  Primary sarcoma: Low FCH uptake | 1

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | 18F-fluoromethylcholine PET/CT
All-Cause Mortality (participants affected / at risk) | 2/64
Serious Adverse Events (participants affected / at risk) | 2/64
Other Adverse Events (participants affected / at risk) | 0/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 18F-fluoromethylcholine PET/CT (N=64)
death within 30 days (Surgical and medical procedures) | 2 (2) — death within 30 days, unrelated to study intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-08-18): https://cdn.clinicaltrials.gov/large-docs/30/NCT01395030/Prot_000.pdf
  • Statistical Analysis Plan (2011-07-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT01395030/SAP_001.pdf